CLINICAL TRIAL: NCT05645991
Title: Effects of Novel Coconut Inflorescence Sap (CSP; COCOZEN) on Age-related Cardiovascular Function
Brief Title: Coconut Sugar Lowers Blood Pressure and Arterial Stiffness in Middle-aged and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Principal Investigator, Brad Fleenor, Associate Professor, Ball State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: COCOZEN
Record Dates: First submitted 2022-11-18; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Aging; Blood Pressure; Arterial Stiffness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Capsules containing aspartame (1.5 g/day) were taken orally once daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo
- Coconut Sap Powder (Experimental): Capsules containing coconut sap powder (CSP; 1.5 g/day) were taken orally once daily for 8 weeks.
  Interventions: Dietary Supplement: Coconut Sap Powder (CSP)

INTERVENTIONS:
Dietary Supplement: Coconut Sap Powder (CSP) — CSP was given once daily (1.5 g/day) for 8 weeks.
  Other Names: COCOZEN; Coconut Inflorescence Sap
  Arms: Coconut Sap Powder
Dietary Supplement: Placebo — Capsules containing aspartame (1.5 g/day) were taken orally once daily for 8 weeks.
  Arms: Placebo

SUMMARY:
The goal of this intervention is to determine the efficacy of coconut sap powder (CSP) to lower arterial stiffness and blood pressure in middle-aged and older adults. Participants will be randomized to the CSP arm or Placebo arm of the study. Primary endpoints include: aortic stiffness assessed by carotid-femoral pulse wave velocity, resting brachial and (non-invasive) carotid blood pressure, and carotid stiffness (e.g. Beta stiffness index, Carotid compliance, Elastic modulus, Distensibility).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18-35 kg/m2
* Brachial blood pressure <140/90
* Nonsmoker
* No known clinical disease, or suggestive signs or symptoms of clinical disease
* Free of alcohol or drug dependence

Exclusion Criteria:

* taking any anti-hypertensive, lipid lowering or other cardiovascular altering medications
* Known allergies to coconut or tree nuts (i.e., cashews, almonds, or pistachios)
* Engaging in vigorous intensity exercise

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Change in aortic stiffness | Baseline and 8 weeks
  Carotid-femoral pulse wave velocity (meters/second)
Change in systolic and diastolic brachial blood pressure | Baseline and 8 weeks
  Manual sphygmomanometer (mmHg)
Change in carotid systolic and diastolic blood pressure | Baseline and 8 weeks
  Applanation tonometry of carotid artery (mmHg)
Change in carotid artery stiffness - beta stiffness index | Baseline and 8 weeks
  Carotid artery Beta stiffness index (AU)
Change in carotid artery stiffness - carotid compliance | Baseline and 8 weeks
  Carotid artery carotid compliance (mmHg/mm^2)
Change in carotid artery stiffness - elastic modulus | Baseline and 8 weeks
  Carotid artery elastic modulus (kilopascals, kPa)
Change in carotid artery stiffness - Young's modulus | Baseline and 8 weeks
  Carotid artery Young's modulus (kilopascals, kPa)
Change in carotid artery stiffness - distensibility | Baseline and 8 weeks
  Carotid artery distensibility (10^-3/kilopascals)

SECONDARY OUTCOMES:
Change in inflammatory biomarker - interleukin 6 | Baseline and 8 weeks
  Biomarker: Interleukin 6 pg/mL
Change in inflammatory biomarker - interleukin 10 | Baseline and 8 weeks
  Biomarker: Interleukin 10 pg/mL
Change in inflammatory biomarker - interleukin 1 beta | Baseline and 8 weeks
  Biomarker: Interleukin 1 beta pg/mL
Change in inflammatory biomarker - tumor necrosis factor alpha | Baseline and 8 weeks
  Biomarker: Tumor necrosis factor alpha pg/mL
Change in inflammatory biomarker - monocyte chemoattractant protein 1 | Baseline and 8 weeks
  Biomarker: Monocyte chemoattractant protein 1 pg/mL
Change in inflammatory biomarker - high sensitivity C-reactive protein | Baseline and 8 weeks
  Biomarker: High sensitivity C-reactive protein mg/mL
Change in oxidative stress biomarkers - superoxide dismutase | Baseline and 8 weeks
  Biomarker: Superoxide dismutase U/mL
Change in oxidative stress biomarkers - Catalase | Baseline and 8 weeks
  Biomarker: Catalase U/mL
Change in oxidative stress biomarkers - Oxidized low density lipoprotein | Baseline and 8 weeks
  Biomarker: Oxidized Low density lipoprotein mU/L

CONTACTS AND LOCATIONS:
Locations (1):
- Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No